CLINICAL TRIAL: NCT02870114
Title: Sociodemographic, Clinic and Psychosocial Aspects of People With Haemophilia in Portugal: a National Survey
Brief Title: National Survey of People With Haemophilia in Portugal
Status: Completed | Type: Observational
Sponsor: University of Minho (Other)
Collaborators: Hospital Sao Joao (Other); Portuguese hemophilia association and other congenital coagulopathies (Unknown)
Responsible Party: Principal Investigator, Patrícia Ribeiro Pinto, Post-doctoral fellow, University of Minho
Other Study IDs: 520101.ID1825
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Haemophilia
Keywords: Haemophilia; Quality of Life; Distress; Hemarthrosis; Pain
MeSH Terms: conditions — Hemophilia A; Hemarthrosis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to implement a national survey to collect information regarding Portuguese people with haemophilia (PWH) on socio-demographic, clinical and psychosocial factors.

DETAILED DESCRIPTION:
This is a cross-sectional design investigation focused on the socio-demographic, clinical and psychosocial characterization of Portuguese people with haemophilia (PWH). All PWH, registered in the Portuguese Hemophilia Association (APH) will be identified in APH registries and contacted through mail, in order to be invited to participate in the first Portuguese survey on haemophilia. In case of acceptance, patients must sign the Informed Consent, fill in the questionnaires and send both back to the investigation team through a pre-paid envelope in the national mail system.

PWH of all ages are invited to participate in this survey. Adults (aged 18 and over) and children/youth from 10 to 17 will answer the questionnaires by self report. Parents of small children (0 to 9) will fill in the proxy versions. All questionnaires are adapted for the specific age groups.

This study will comply with ethic guidelines and was approved by the Life Sciences and Health Ethics Subcommittee (University of Minho) and is registered on the Portuguese authority for data collection (CNPD).

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A or B
* Portuguese nationality

Exclusion Criteria:

* Acquired Haemophilia
* Psychiatric or neurological deficit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with Haemophilia A or B, of any age and gender, registered in the Portuguese Haemophilia Association
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life in Adults as assessed by A36Hemofilia-Qol | 1 year
Health Related Quality of Life in Children as assessed by Canadian Haemophilia Outcomes-Kids Life Assessment Tool | 1 year
  Health Related Quality of Life in Children
Pain Intensity | 1 year
  Pain Questionnaire developed specifically for this investigation to assess PWH (based on Wallny's Pain Questionnaire for PWH and Brief Pain Inventory).
Pain Location | 1 year
  Pain Questionnaire developed specifically for this investigation to assess PWH (based on Wallny's Pain Questionnaire for PWH and Brief Pain Inventory).
Pain Duration | 1 year
  Pain Questionnaire developed specifically for this investigation to assess PWH (based on Wallny's Pain Questionnaire for PWH and Brief Pain Inventory).

SECONDARY OUTCOMES:
Total score of Haemophilia-related functional limitations as assessed by Haemophilia Activities List (HAL) and Pediatric HAL | 1 year
Anxiety score as assessed by PROMIS-Anxiety Short Form v1.0 | 1 week
  Assessmet of Anxiety
Depression score as assessed by PROMIS-Depression Short Form v1.0 | 1 week
Illness Perception as assessed by IPQ-R | 1 year
Pain Catastrophizing as assessed by CSQ - Catastrophizing Subscale | 1 year
Number of Joint Bleeds | 1 year
Presence of inibitors | 1 year
Number of target joints | 1 year
Type of sports practiced by PWH | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia R Pinto, PhD, Principal Investigator — Life and Health Sciences Research Institute
Locations (1):
- Life and Health Sciences Research Institute, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No